CLINICAL TRIAL: NCT04750005
Title: Twelve Week Clinical Efficacy of Virtually Supervised Mouth Rinse and Flossing: Effect on Plaque and Gingivitis
Brief Title: A Twelve Week Study of Virtually Supervised Mouth Rinse and Flossing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CCSORC002906; CCSORC002906 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — American Dental Association

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brush only Group (Active Comparator): Participants assigned to this group will brush their teeth using soft bristled toothbrush and colgate cavity protection toothpaste as directed under virtual supervision once daily during the week. Participants will brush second time unsupervised daily in the evening and twice daily over the weekend/holidays at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Ref Toothbrush
- Brush/Rinse Group (Experimental): Participants assigned to this group will perform their regimen (brushing [soft bristled toothbrush and colgate cavity protection toothpaste] and rinsing [listerine cool mint antiseptic mouthwash]) as directed under virtual supervision once daily during the week. Participants will brush and rinse a second time unsupervised daily in the evening at home. At home, participants will brush and rinse a second time unsupervised daily in the evening and twice daily over the weekend/holidays. First product use will occur at the site under supervision.
  Interventions: Other: Listerine Cool Mint; Other: Colgate Cavity Protection Toothpaste; Other: American Dental Association (ADA) Ref Toothbrush
- Brush/Floss Group (Experimental): Participants assigned to this group will perform their regimen (brushing and flossing) as directed under virtual supervision once daily during the week. At home, participants will brush a second time unsupervised daily in the evening. Over the weekend and holidays, participants will brush and floss once daily. Only brushing will be performed a second time in the evening. First product use will occur at the site under supervision.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: Reach Unflavored Waxed Dental Floss; Other: American Dental Association (ADA) Ref Toothbrush
- Brush/Floss/Rinse Group (Experimental): Participants assigned to this group will perform their regimen (brushing [soft bristled toothbrush and colgate cavity protection toothpaste], flossing [reach unflavored waxed dental floss] and rinsing [listerine cool mint antiseptic mouthwash]) as directed under virtual supervision once daily during the week. Participants will brush and rinse a second time unsupervised daily in the evening. Over the weekend and holidays, participants will brush, floss and rinse once daily. Only brushing and rinsing will be performed a second time in the evening at home.
  Interventions: Other: Listerine Cool Mint; Other: Colgate Cavity Protection Toothpaste; Other: Reach Unflavored Waxed Dental Floss; Other: American Dental Association (ADA) Ref Toothbrush

INTERVENTIONS:
Other: Listerine Cool Mint — Participants use 20 mL of Listerine cool mint mouth rinse for 30 sec after brushing twice a day.
  Arms: Brush/Floss/Rinse Group; Brush/Rinse Group
Other: Colgate Cavity Protection Toothpaste — Participants used Colgate cavity protection toothpaste for brushing teeth twice daily.
Other: Reach Unflavored Waxed Dental Floss — Participants after brushing for 1 minute, rinse mouth with water and FLOSS once a day in first use.
  Arms: Brush/Floss Group; Brush/Floss/Rinse Group
Other: American Dental Association (ADA) Ref Toothbrush — Participants will brush twice daily for 1 minute with the toothpaste and soft bristled toothbrush provided.

SUMMARY:
The purpose of this study is to evaluate the efficacy of brushing, flossing, and rinsing with an alcohol containing essential oil mouth rinse; brushing and flossing; versus brushing and rinsing with an alcohol containing essential oil mouth rinse; and brushing only for the prevention and reduction of plaque and gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand (participants capable of reading the documents)
* Adequate oral hygiene (that is brush teeth daily and exhibit no signs of oral neglect)
* Negative pregnancy urine tests (females of childbearing potential only)
* Females of childbearing potential must be using a medically-acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the study
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* A minimum of 10 percent (%) bleeding sites based on the expanded bleeding index (BI)
* Participants will have evidence of some gingivitis; there will be no minimum or maximum mean MGI score for gingivitis or TPI score for plaque; mild to severe gingivitis and mild to moderate periodontitis
* No more than 3 sites having pocket depths of 5 millimeter (mm) and no sites that are greater than 5 mm in depth

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses and red food dye; Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients (or other ingredients in the products)
* Dental prophylaxis within four weeks prior to Screening/Baseline visit
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Use of antibiotics, anti-inflammatory or anticoagulant therapy during the study or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the investigator
* Suspected alcohol or substance abuse (example., amphetamines, benzodiazepines, cocaine, marijuana, opiates

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Whole-mouth Mean Modified Gingival Index (MGI) Score After 12 Weeks of Product use | 12 Weeks
  Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Mean Turesky Plaque Index (TPI) Score After 12 Weeks of Product use | 12 Weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).

SECONDARY OUTCOMES:
Marginal and Interproximal Mean Turesky Plaque Index (TPI) Score After 4 and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).
Marginal and Interproximal Mean Modified Gingival Index (MGI) Score After 4 and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Marginal Mean Expanded Bleeding Index (EBI) Score After 4 and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Whole-mouth Mean Turesky Plaque Index (TPI) Score After 4 Weeks of Product use | 4 Weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).
Whole-mouth Mean Modified Gingival Index (MGI) Score After 4 Weeks of Product use | 4 Weeks
  Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-mouth and Interproximal Mean Bleeding Index (BI) After 4 and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Whole-mouth and Interproximal Percent Bleeding Sites, Based on the EBI Score After 4 and 12 Weeks of Product use | 4 Weeks and 12 Weeks
  Percent bleeding sites will be calculated by taking the total number of sites with bleeding score greater than 0 divided by the total number of sites assessed for each participant. Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Interproximal of the Proximal Marginal Plaque Index Score After 4 and 12 Weeks | 4 Weeks and 12 Weeks
  Interproximal Plaque area will be assessed using the PMI on the facial and lingual surfaces. Distal proximal and mesial proximal will be assessed on all teeth including the distal of the second molar using the following scoring system: 0 = No plaque;
  1 = Separate flecks of plaque covering less than 1/3 of the area; 2 = Discrete areas or bands of plaque covering less than 1/3 of the area; 3 = Plaque covering 1/3 of the area; 4 = Plaque covering more than 1/3 but less than 2/3 of the area; 5 = Plaque covering 2/3 or more of the area.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Rich SK, Friedman JA, Schultz LA. Effects of flossing on plaque and gingivitis in third grade schoolchildren. J Public Health Dent. 1989 Spring;49(2):73-7. doi: 10.1111/j.1752-7325.1989.tb02029.x. PMID 2709366
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] CHILTON NW. Studies in the design and analysis of dental experiments. II. A four-way analysis of variance. J Dent Res. 1960 Mar-Apr;39:344-60. doi: 10.1177/00220345600390021601. No abstract available. PMID 13809868
- [Background] Saxton CA, van der Ouderaa FJ. The effect of a dentifrice containing zinc citrate and Triclosan on developing gingivitis. J Periodontal Res. 1989 Jan;24(1):75-80. doi: 10.1111/j.1600-0765.1989.tb00860.x. PMID 2524573
- [Background] Van der Weijden GA, Timmerman MF, Nijboer A, Reijerse E, Van der Velden U. Comparison of different approaches to assess bleeding on probing as indicators of gingivitis. J Clin Periodontol. 1994 Oct;21(9):589-94. doi: 10.1111/j.1600-051x.1994.tb00748.x. PMID 7806674
- [Background] Benson BJ, Henyon G, Grossman E. Clinical plaque removal efficacy of three toothbrushes. J Clin Dent. 1993;4(1):21-5. PMID 8357508
- [Background] Newman, MG, Takei, H, Klokkevold, PR, Carranza, FA; 2018; Newman and Carranza's Clinical Periodontology E-Book, 13th Edition; Saunders; p.387.
- [Background] Sharma NC, Charles CH, Qaqish JG, Galustians HJ, Zhao Q, Kumar LD. Comparative effectiveness of an essential oil mouthrinse and dental floss in controlling interproximal gingivitis and plaque. Am J Dent. 2002 Dec;15(6):351-5. PMID 12691269
- [Background] Sharma N, Charles CH, Lynch MC, Qaqish J, McGuire JA, Galustians JG, Kumar LD. Adjunctive benefit of an essential oil-containing mouthrinse in reducing plaque and gingivitis in patients who brush and floss regularly: a six-month study. J Am Dent Assoc. 2004 Apr;135(4):496-504. doi: 10.14219/jada.archive.2004.0217. PMID 15127875
- [Background] Bauroth K, Charles CH, Mankodi SM, Simmons K, Zhao Q, Kumar LD. The efficacy of an essential oil antiseptic mouthrinse vs. dental floss in controlling interproximal gingivitis: a comparative study. J Am Dent Assoc. 2003 Mar;134(3):359-65. doi: 10.14219/jada.archive.2003.0167. PMID 12699051
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC002906&attachmentIdentifier=b846a7b2-b2c9-4957-a4be-a768894a56ba&fileName=CCSORC002906_Summary_CSR___Redacted.pdf&versionIdentifier=